CLINICAL TRIAL: NCT06396156
Title: Anterior Chamber Versus Retropupillary Iris-claw Intraocular Lens Fixation in Aphakic Children With Insufficient Capsular Support.
Brief Title: Anterior Versus Posterior Artisan Intraocular Lens Fixation in Aphakic Children With Insufficient Capsular Support.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Awadein, Professor of Ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-45-2022
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cataracts Infantile; Subluxation of Lens; Intraocular Lens Complication; Corneal Endothelial Cell Loss
Keywords: aphakia; subluxation; corneal endothelium; iris-claw lens
MeSH Terms: conditions — Lens Subluxation; Corneal Endothelial Cell Loss; Aphakia; Joint Dislocations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- anterior chamber iris-claw lens (Active Comparator): Eyes that receive Artisan IOL that is fixed anterior to the iris
  Interventions: Procedure: Anterior enclavation
- Retro-pupillary Iris- Claw lens (Active Comparator): Eyes that receive Artisan IOL that is fixed posterior to the iris
  Interventions: Procedure: Posterior enclavation

INTERVENTIONS:
Procedure: Anterior enclavation — Anterior enclavation of iris-claw lens
  Arms: anterior chamber iris-claw lens
Procedure: Posterior enclavation — Posterior enclavation of iris-claw lens
  Arms: Retro-pupillary Iris- Claw lens

SUMMARY:
The Artisan lens (Artisan Aphakic, Ophtec BV) is an iris- claw lens designed for implantation in children with insufficient capsular support. In spite of less surgical manipulations and a relatively shorter operation time, the procedure carries the risk of corneal endothelial cell loss or dis-enclavation, particularly in children. However, most of the studies that studied iris-claw lenses in aphakic children were retrospective evaluated only a single technique; either anterior or retropupillary fixation, or comparable to other techniques of fixation. Thus the aim of this work is to prospectively compare the 2 techniques of iris-claw lens implantation and their effects on central endothelial cell density, the anatomical and visual outcome, as well as the complications' rate.

DETAILED DESCRIPTION:
Children for the study will be recruited from the Pediatric Ophthalmology Clinics in Cairo University Hospitals. Children will be included if they have aphakia with insufficient capsular support, hereditary lens subluxation. microspherophakia . or traumatic lens subluxation > 180 degrees that requires lensectomy and intraocular lens implantation .

Patients recruited for this study will be assigned into 2 groups:

1. Group A: will have implantation of an anterior chamber iris-claw lens (Ophtec BV, Groningen, The Netherlands)
2. Group B: Wil have implantation of a retropupillary iris-claw lens (Ophtec BV, Groningen, The Netherlands)

Preoperative Evaluation

Demographics and History Taking Baseline demographic data will be collected from all patients including

1. Age at time of surgery
2. Gender
3. Laterality
4. History of trauma
5. History of any previous ocular interventions.

   Systemic Workup:

   Patients without evidence of trauma had a complete workup in conjunction with a pediatrician for the underlying cause of subluxation or absent capsular support

   Ocular Examination:
   * Measurement of best-corrected visual (BCVA) using the tumbling E chart or the Allen's picture chart will be done. Visual acuity will be expressed as logMAR acuity
   * Detailed slit lamp examination:

   Evaluation of the cornea for clarity and regularity Evaluation of the anterior chamber Evaluation of the iris for - Iris structure and iris defects - Tremulousness

   - Sphincteric ruptures and traumatic injuries to the iris including iridodialysis, atrophy, and traumatic aniridia

   - Synechiae between the iris and the lens/capsular remnants Examination of the pupil for

   - Pupil size undilated and after dilatation

   - Centralization of the pupil Evaluation of the capsular support and any residual lens matter, Sommering ring, or Elschninng pearls in aphakic cases Evaluation of the lens in subluxated cases for

   - Extent of subluxation

   - Direction of subluxation

   - Integrity of the zonules including any elongation or anomalies in the zonules

   - Relation of the lens to the center of the pupil through an undilated and a dilated exam

   - Clarity of the lens

   - Change in the lens position with the supine position

   - Tremulousness' of the lens

   - Dilated fundus examination using both slit lamp biomicroscopy and indirect ophthalmoscopy.

   - Measurement of the IOP using Perkins tonometer (Haag Streit, UK): Measurement of IOP will be done under topical anesthesia in cooperative children and under general anesthesia at the start of surgery in uncooperative children
   * Examination of the angle of anterior chamber using the Swan- Jacob's goniolens under general anesthesia at the start of the surgery.
   * Evaluation of central corneal thickness (CCT) using a handheld pachymeter (DGH55, Exton, USA).

   Evaluation of corneal endothelium:

   Corneal endothelial cell count (ECC) will be evaluated using non-contact Specular Microscope (Konan Medical KSS-300, Inc., Hyogo, Japan) for all children. only sharp images with easily identified cell borders will be analyzed. The endothelial cell density (ECD) will be calculated with center method in all images. Fixed number of cells will be used in all scans to eliminate variability. Manual selection of cells will be performed in all scans. A single island of contiguous cells with well identified borders will be used for calculations.

   Anterior Segment Optical Coherence Tomography (AS-OCT):

   All subject eyes will be scanned with a hand-held anterior segment optical coherence tomography (HH AS-OCT); RTVue RT-100 system (Optovue Inc., Fremont, CA). A non-contact technique will be used for scanning, with the child lying supine without sedation. All scans will be performed with the pupil undilated and under mesopic conditions. each eye will be imaged at least 3 scans per visit.

   Corneal thickness mapping:

   A pachymetry scan pattern, with 6-mm scan diameter and eight radials, will be chosen to map the cornea. The RTVue corneal adapter module software provided the pachymetry map of total corneal thickness, automatically. Central corneal thickness will be automatically calculated in µm as the central distance between the epithelium and endothelium.

   Anterior chamber angle assessment:
   * Image acquisition:

   Scanning of the angle will be performed on the nasal and temporal quadrants at 3 and 9 o'clock under mesopic conditions with the device's software set to Angle mode. In this mode, a 3 x 2.3 mm area centered at the limbus will be analyzed. Each quadrant will be scanned three times, and the investigator will choose the image showing the best quality and least noise.

   - Angle morphology: Identification of the anterior chamber angle structures will be performed. Identification of scleral spur (SS) (The anatomical landmark), trabecular meshwork, Schlemm's canal before surgery.

   Angle abnormalities including abnormal angle membrane, peripheral anterior synechiae (PAS), primary congenital glaucoma (PCG) like changes will be documented in pre and postoperative scans.

   - Anterior chamber angle parameters The anterior chamber (AC) angle width The angle opening distance (AOD) (µm)

   IOL power calculation:

   IOL power calculation will be performed using optical biometry. In uncooperative children and children in whom optical biometry could not be performed, an A-scan biometry will be performed using contact technique. IOL power will be calculated using either SRK-T and Holladay 1 formula. An A constant of 115.7 and 116.8 will be assigned for the anterior chamber and posterior iris-claw lens, respectively. Emmetropia will be targeted in all patients.

   Surgical technique:

   All surgeries will be performed under general anesthesia. In all the eyes that required lensectomy, the procedure will be performed through an anterior corneal approach. A 23-gauge MVR knife will be used to create two side ports at 3 o'clock and 9 o'clock. A cohesive viscoelastic will be injected in retrolenticular space. Then, the MVR blade will be used to create 2 incisions at the equator of the subluxated lens, and slightly widened. A 23-gauge bimanual irrigation and aspiration system will be used to aspirate lens matter. Then a 23-G vitrectomy probe will be used for lens capsule removal. Sweeping of anterior chamber using spatula will be performed to ensure the absence of vitreous strands. Miosis will be achieved by injecting intra-cameral pilocarpine 1% then a peripheral iridectomy at 11 or 1 o'clock will be performed using the vitrector probe. A cohesive viscoelastic will be injected, and then a superior limbal corneal incision of 6 mm will be constructed, but not opened. In Group A, anterior chamber iris claw fixation will be done. The lens will be introduced using the curved Clayman forceps with its vault facing up, and then enclavated at 3 and 9 o'clock positions anterior to the iris. In the retropupillary group (Group B), the IOL will be introduced behind the pupil and enclavated behind the iris. Corneal wounds will be them closed using 10/0 nylon sutures.

   Postoperative regimen:

   Topical steroids and antibiotics will be prescribed for 6-8 weeks after surgery. Topical tropicamide 1% will be prescribed to be used twice per day for 1 week to decrease pigment dispersion. Removal of sutures will be done 6 weeks after surgery.

   Postoperative Follow-Up:

   Patients will be followed up at 1 day, 1 week, 1 month, 6 months, and 12 months after surgery. More frequent follow-up will be performed whenever needed.

<!-- -->

1. Clinical examination:

   All patients will be examined on the first day after surgery for o Corneal clarity o Anterior chamber reaction and pigment dispersion o Stability and centration of the IOL o Patency of the peripheral iridectomy

   o IOP measurement Clinical examination will be then repeated at each follow-up visit
2. Automated refraction or retinoscopy and prescription of spectacles:

   A dilated refraction will be performed 2 weeks after suture removal (8 weeks after surgery), Any residual refractive error will be corrected fully in all patients using single vision glasses. In older children, bifocal spectacles will be prescribed.
3. Measurement of best-corrected visual acuity (BCVA) Measurement of BCVA will be performed after prescription of spectacles, then repeated at 6 and 12 months. Tumbling E chart will be used for literate children. Teller cards will be used in few illiterate children. Children who show interocular difference in the visual acuity ≥ 3 logMAR lines will be prescribed patching to the better seeing eye according to the PEDIG guidelines.
4. Measurement of central endothelial cell density A repeat specular microscopy will be performed at 1 month, 6 months, and 12 months after surgery. Sharp images with easily identified cell borders will be analyzed. Manual center method will be used for cell identification. Fixed number of cells will be used in all analyses.
5. Assessment of changes in central corneal thickness and anterior chamber angle will be performed using hand-held optical coherence tomography (OCT), A repeat anterior segment OCT will be performed at 1 month, 6 months, and 12 months after surgery.
6. Ultrasound biomicroscopy:

UBM scanning (VuMAX HD, Sonomed Escalon, New York) will be performed at the end of 1-year follow-up. Examination will be performed with the patient in the supine position to measure IOL tilt and decentration.

ELIGIBILITY:
Inclusion Criteria:

* Hereditary lens subluxation that requires lensectomy and intraocular lens implantation.
* Traumatic lens subluxation that requires lensectomy and intraocular lens implantation.
* Microspherophakia that requires lensectomy and intraocular lens implantati
* Aphakia with insufficient capsular support.

Exclusion Criteria:

* Preoperative central endothelial cell density (CECD) less than 2500 cells/mm2
* Preoperative anterior chamber depth (ACD) less than 3 mm.
* Severely damaged iris.
* History of uveitis or glaucoma.
* Macular lesions or previous retinal surgery

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Endothelial cell loss | 1 year
  Percentage of endothelial cell loss from the baseline value

SECONDARY OUTCOMES:
Best-corrected visual acuity | 1 year
  Best-corrected distance log-MAR visual acuity
Anterior chamber angle | 1 year
  Width of anterior chamber angle by OCT
Intraocular pressure | 1 year
  Measured intraocular pressure by applanation
IOL tilt | 1 year
  Degree of tilt of intraocular lens measured by UBM
IOL decentration | 1 year
  Degree of decentration of lens measured by UBM

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Saeed, MD, Study Chair — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University Pediatric Hospital, Cairo
  - Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gawdat GI, Taher SG, Salama MM, Ali AA. Evaluation of Artisan aphakic intraocular lens in cases of pediatric aphakia with insufficient capsular support. J AAPOS. 2015 Jun;19(3):242-6. doi: 10.1016/j.jaapos.2015.03.014. PMID 26059670
- [Background] Yulia DE, Barliana JD, Soeharto DA. Visual outcome of intraocular Iris-Claw lens implantation in Indonesian children with ectopia lentis. Taiwan J Ophthalmol. 2022 Feb 28;13(3):335-340. doi: 10.4103/tjo.tjo_58_21. eCollection 2023 Jul-Sep. PMID 38089522
- [Background] Cevik SG, Cevik MO, Ozmen AT. Iris-claw intraocular lens implantation in children with ectopia lentis. Arq Bras Oftalmol. 2017 Mar-Apr;80(2):114-117. doi: 10.5935/0004-2749.20170027. PMID 28591285
- [Background] Yulia DE, Soeharto DA. Efficacy and Safety of Iris-Claw Intraocular Lens in Pediatric Ectopia Lentis: A Literature Review. J Curr Ophthalmol. 2023 Aug 11;35(1):1-10. doi: 10.4103/joco.joco_249_22. eCollection 2023 Jan-Mar. PMID 37680281